CLINICAL TRIAL: NCT00812604
Title: Effect of an Analgesic Ointment on the Relief of Temporomandibular Joint and Masticatory Muscle Pain: a Randomized, Double Blinded, Placebo-controlled Study.
Brief Title: Analgesic Ointment on Temporomandibular Joint and Masticatory Muscle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Wing Kit, Ricky, Associate Professor, Orthodontics, Faculty of Dentistry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKCTR-466
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-05

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ping On Ointment (Experimental): Ping On Ointment
  Interventions: Drug: Ping On Ointment
- Vaseline (Placebo Comparator): Vaseline with minor trace of Ping On ointment to give medicinal smell
  Interventions: Drug: Vaseline

INTERVENTIONS:
Drug: Ping On Ointment — Ping On Ointment
  Other Names: TCM topical analgesic
  Arms: Ping On Ointment
Drug: Vaseline — Placebo
  Arms: Vaseline

SUMMARY:
The purpose of this study is to compare the effectiveness of using topical cream of Ping On Ointment and using Vaseline cream in the treatment of temporomandibular joint (TMJ) and masticatory muscle pain, in order to establish the true efficacy of Ping On Ointment. Both Ping On Ointment and Vaseline are considered intervention.

DETAILED DESCRIPTION:
Aims: To compare the effectiveness of using topical cream of Ping On Ointment and using Vaseline cream in the treatment of temporomandibular joint (TMJ) and masticatory muscle pain, in order to establish the true efficacy of Ping On Ointment. Methods: In this randomized, double-blinded, placebo-controlled trial, 55 subjects with TMJ and/or masticatory pain (Group 1 patients according to the Research Diagnostic Criteria for Temporomandibular Disorder (RDC/TMD) received Ping On Ointment for 4 weeks; or placebo for 4 weeks. Subjects were evaluated with standard measures of efficacy: pain intensity measured by visual analogue scale and maximal comfortable mandibular opening, at baseline and again after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Self report of facial ache or pain in the muscles of mastication, the TMJ, or the region in front of ear or inside the ear
2. Positive clinical diagnosis of TMDs. The TMD diagnosis is classified using axis I of the research diagnostic criteria ( RDC) for TMDs. The RDC diagnosis consists of joint pain at rest ( spontaneous pain) and evoked pain (hyperalgesia) on palpation of the TMJ, TMJ reduction consists of reciprocal clicking or joint noise with mandibular movement examination.
3. For joint pain complaint, subjects will be required to have a self-report of at least 1 month of daily or nearly-daily pain.
4. Subjects with myogenic pain will be included if they meet inclusion and exclusion criteria since patients with TMDs are known to exhibit muscle pain secondary to their joint dysfunction.

Exclusion Criteria:

1. Subjects with infectious arthritis, crystal induced arthropathies, musculoskeletal disorders, subjects with a primary diagnosis of myofascial pain based on the RDC;
2. Subjects with pain attributable to confirmed migraine or head pain condition other than tension headache;
3. Subjects with acute infection or other significant disease of teeth, ears, eyes, nose or throats; subjects with untreated depressive disorder or not on stable antidepressant medication for more than 6 months;
4. Subjects with dental diseases that required ongoing treatment, which would confound the evaluation of orofacial pain;
5. Subjects who are not competent in giving consents.
6. Pregnant or lactating women
7. Subjects with sensitivity to the ingredient of Ping On Ointment will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricky W. K. Wong, PhD, Principal Investigator — Orthodontics, Faculty of Dentistry, University of Hong Kong
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Li LC, Wong RW, Rabie AB. Clinical effect of a topical herbal ointment on pain in temporomandibular disorders: a randomized placebo-controlled trial. J Altern Complement Med. 2009 Dec;15(12):1311-7. doi: 10.1089/acm.2009.0129. PMID 20001836

RESULTS

PARTICIPANT FLOW:
Groups:
- Ping On Ointment Group: Ping On Ointment was used
- Placebo Group: Vaseline with minor trace of Ping On Ointment was used
Period: Overall Study
Arm/Group | Ping On Ointment Group | Placebo Group
Started | 28 | 27
Completed | 23 | 22
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ping On Ointment Group | Placebo Group | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.14 (9.296) | 43.96 (13.127) | 45.51 (11.401)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  Hong Kong | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy in the Treatment of TMJ and Muscle Pain
Description: The efficacy in the treatment of TMJ and muscle pain is measured by a visual analogue scale (VAS).
  The VAS consists of a 100 mm line, anchored with the extremes of pain intensity represented as "no pain" ( 0 mm) and " worst pain possible" ( 100 mm).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ping On Ointment Group | Placebo Group
Number analyzed (Participants) | 23 | 22
units on a scale | 21.93 (18.07) | 40.81 (14.44)

2. Secondary Outcome: The Mandibular Function.
Description: The mandibular function, the maximal comfortable mandibular opening measured in millimeters at the subjects's maximum incisor to incisor mouth opening using a ruler.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ping On Ointment Group | Placebo Group
Number analyzed (Participants) | 23 | 22
mm | 4.435 (6.680) | 0.818 (3.404)

ADVERSE EVENTS:
Arm/Group | Ping On Ointment Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

LIMITATIONS AND CAVEATS:
In this study, the subjects were screened by clinical examinations and self-reported questionnaires. Ideally, the diagnosis should be made with a combination of radiographs, Magnetic Resonance Imaging or Computer Tomography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes